CLINICAL TRIAL: NCT04810910
Title: Clinical Study of a Personalized Neoantigen Vaccine in Pancreatic Cancer Patients Following Surgical Resection and Adjuvant Chemotherapy
Brief Title: Personalized Neoantigen Vaccine in Pancreatic Cancer Patients Following Surgical Resection and Adjuvant Chemotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: Hangzhou Neoantigen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Liu Yang, MD, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INEO-P-005
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Resectable Pancreatic Cancer
MeSH Terms: interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Adjuvants, Immunologic; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized neoantigen vaccines (Experimental): iNeo-Vac-P01 (peptides)： 4 x 300 mcg per peptide given on days 1, 4, 8, 15, 22, 52, and 82 for a total of 7 doses;
  GM-CSF: 4 x 40 mcg (total dose 160 mcg) given on days 1, 4, 8, 15, 22, 52, and 82 for a total of 7 doses
  Interventions: Biological: iNeo-Vac-P01; Other: GM-CSF

INTERVENTIONS:
Biological: iNeo-Vac-P01 — iNeo-Vac-P01 (peptides)： 300 mcg per peptide
  Other Names: Neoantigen peptides
Other: GM-CSF — GM-CSF: 40 mcg
  Other Names: immune adjuvant; granulocyte-macrophage colony stimulating factor

SUMMARY:
This research study is evaluating a new type of pancreatic cancer vaccine called "Personalized Neoantigen Cancer Vaccine" as a possible treatment for pancreatic cancer patients following surgical resection and adjuvant chemotherapy. The purpose of the clinical study is evaluating the safety, tolerability and partial efficacy of the personalized neoantigen cancer vaccine in the treatment of resectable pancreatic cancer, so as to provide a new personalized therapeutic strategy.

It is known that cancer patients have mutations (changes in genetic material) that are specific to an individual patient and tumor. These mutations can cause the tumor cells to produce proteins that appear very different from the body's own cells. It is possible that these proteins used in a vaccine may induce strong immune responses, which may help the participant's body fight any tumor cells that could cause the cancer to come back in the future. The study will examine the safety of the vaccine when given at several different time points and will examine the participant's blood cells for signs that the vaccine induced an immune response.

ELIGIBILITY:
Inclusion Criteria：

1. Must freely sign informed consent;
2. Aged 18 to 70 years old;
3. Histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma;
4. Must provide all exons of tumor tissue sequencing data, transcriptome sequencing data and the peripheral blood of all exons sequencing data;
5. ECOG score is 0 or 1;
6. Completed an R0 or R1 surgical resection as determined by pathology；
7. Completion of at least 4 months of adjuvant chemotherapy with ticgio monotherapy or mFOLFIRINOX;
8. Completion of imaging records 1 week before personalized immunotherapy, including but not limited to full-body PET-CT and brain MRI,
9. The end of chemotherapy is followed by a one-week natural washout period；
10. Haematological index：

    * White blood cells ≥ 3500 / MCL
    * Lymphocytes > 800/ MCL
    * neutrophils > 1500/ MCL
    * Platelets > 100000 / MCL
    * Hemoglobin >10.0g/dL
    * Total serum bilirubin <1.5× upper limit of normal value (ULN)
    * AST/ALT<2.0 times the upper limit of normal
    * Serum creatinine <1.5 times the upper limit of normal；
11. Pregnant, lactating women and women of child-bearing age must have a negative pregnancy test within 7 days before entering the group, and short-term have no fertility plan, and are willing to take protective measures (contraception or other birth control methods) before and during the clinical trial;
12. Good compliance, able to follow research protocols and follow-up procedures.

Exclusion Criteria:

1. Evidence of disease recurrence or metastasis following surgical resection at any time prior to the first vaccination administration.
2. Diagnosed as other malignant tumor;
3. No neoantigen was found in the sequencing data;
4. There have been bone marrow or stem cell transplants;
5. Received systemic glucocorticoids with immunosuppressants;
6. Received other polypeptide inoculation 4 weeks before treatment; Patients may not be vaccinated with other polypeptides 8 weeks after the last individualized tumor targeted polypeptides trentment;
7. With HIV, HCV, HBV infection, severe asthma, autoimmune disease, immunodeficiency or treated with immunosuppressive drugs;
8. Uncontrolled complications include, but are not limited to, active infection, symptomatic congestive heart failure, unstable angina pectoris, and arrhythmias;
9. Infected with herpes virus (except those with scabs of more than 4 weeks)；
10. Infected with respiratory virus (except those who have recovered for more than 4 weeks);
11. Have severe coronary or cerebrovascular disease, or other conditions considered ineligible by the investigator;
12. Drug abuse. Clinical, psychological or social factor result in affecting informed consent or research implementation;
13. Have a history of drug or polypeptide allergies, or people who are allergic to other potential immunotherapies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing clinical and laboratory adverse events (AEs) | 1 years
  Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v5.0
Relapse Free Survival(RFS) | 4 years
  Time from surgery to any recurrence

SECONDARY OUTCOMES:
Overall Survival(OS) | 4 years
  Time from surgery to death or last follow-up

OTHER OUTCOMES:
Measurement of CD4/CD8 T lymphocyte subsets | 2 years
The polypeptide antigen - induced IFN-γ T cells responses | 2 years
Peripheral blood T cell receptor sequencing analysis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yang Liu, Liu, Principal Investigator — Zhejiang Provincial People's Hospital
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No